CLINICAL TRIAL: NCT03771742
Title: Randomized Prospective Study to Evaluate Cranial Dermatomal Spread of Modified Paramedic Sagittal Versus Transverse Approach TMQLB for Adrenal Surgery
Brief Title: Modified Paramedic Sagittal vs. Transverse TMQLB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Cui Xulei, Attending physician, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: cuixule6
Record Dates: First submitted 2018-12-09; First posted 2018-12-11 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Nerve Block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transverse TMQLB (Active Comparator): Patients in this group will receive the transmuscular quadratus lumborum block before surgery using the transverse scan, in-plain, posterior to anterior approach. 0.6ml 0.375% ropivocaine was injected when the correct needle location is confirmed.
  Interventions: Procedure: transverse scan, in-plane, posterior-anterior TMQLB
- paramedian sagittal TMQLB (Experimental): Patients in this group will receive the transmuscular quadratus lumborum block before surgery using the para-sagittal scan, in-plain, caudal to cephalic approach.0.6ml 0.375% ropivocaine was injected when the correct needle location is confirmed.
  Interventions: Procedure: paramedian sagittal scan, in-plane, caudal-cranial TMQLB

INTERVENTIONS:
Procedure: transverse scan, in-plane, posterior-anterior TMQLB — The patients will receive the transmuscular quadratus lumborum block(TMQLB) before surgery using the transverse scan, in-plain, posterior to anterior approach. 0.6ml/kg 0.375% ropivocaine is injected when the correct needle location is confirmed.
  Arms: transverse TMQLB
Procedure: paramedian sagittal scan, in-plane, caudal-cranial TMQLB — The patients will receive the transmuscular quadratus lumborum block(TMQLB) before surgery using the paramedic sagittal scan, in-plain, caudal-cephalic approach.0.6ml/kg 0.375% ropivocaine is injected when the correct needle location is confirmed.
  Arms: paramedian sagittal TMQLB

SUMMARY:
The classical transmuscular qudratus lumborum block(TMQLB) described by Borglum aims to provide lower thoracic paravertebral space(PVS) and sympathetic blockade by injecting local anesthetics between QL and PM muscle at the L3-L4 vertebral level using a transverse scan, posterior-anterior, in-plane approach. Recently, a paramedian sagittal oblique(TMQLB) approach has been introduced to facilitate cranial spread by injecting the local in a caudal to cranial direction. Currently, there are no data comparing the two techniques mentioned above with regards to extent of spread for PVS. Our objective is to investigate the extent of cranial dermatomal spread of TMQLB when equal dosage(ml/kg) of local anesthetic are injected with the transverse versus an modified paramedian sagittal approach for patients undergoing laparoscopic adrenalectomy. In addition, the investigators wish to compare the performance time, caudal dermatomal spread of TMQLB and postoperative analgesia effect.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 yrs
* American Society of Anesthesiologists physical statusⅠ-Ⅲ
* Undergo laparoscopic adrenalectomy
* Informed consent
* Able to cooperate with study process

Exclusion Criteria:

* Allergy to local anesthetic and other medications used in the study
* Patient refusal or lack of informed consent
* Coexisting hematological disorder or with deranged coagulation parameters
* Pre-existing major organ dysfunction such as hepatic and renal failure
* History of previous renal surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-17 (Actual)

PRIMARY OUTCOMES:
Cephalic sensory dermatomal spread | 20 minutes after block performance

SECONDARY OUTCOMES:
Time to performance of procedure | Duration of procedure
Total sensory dermatomal spread | 20 minutes after block performance
Incidence of complication | Within 48hours after surgery
Caudal sensory dermatomal spread | 20 minutes after block performance
cumulative rate of rescue analgesics usage | At 0,2,4,8,12,24,48 hours after surgery
NRS pain scores | At 0,2,4,8,12,24,48hours after surgery
  patients will evaluate their pain intensity with the numerical rating scale (NRS), where 0 indicates no pain, and 10 indicates the most severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Xulei CUI, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China